CLINICAL TRIAL: NCT00895856
Title: Evaluation of the Functional Capacity in Institutionalized Elders Who Do Not Receive Physiotherapic Assistance
Brief Title: Functional Capacity in Institutionalized Elders
Status: Completed | Type: Observational
Sponsor: Centro de Estudos Superiores de Maceio (Other)
Responsible Party: Juliana Fonseca Pontes, CESMAC - Centro de Estudos Superiores de Maceió
Other Study IDs: CEP - 414/2008
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2009-05-11 (Estimated); Status verified 2009-05

CONDITIONS: Elderly
Keywords: Physiotherapy; Aged; Functionality; Physiotherapic assistance; Functional capacity
MeSH Terms: interventions — Aging

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Old-aged people
  Interventions: Other: Evaluation of the functional capacity

INTERVENTIONS:
Other: Evaluation of the functional capacity — An evaluation (questionnaire) was performed by the Katz Index of individuals in this group, including personal issues (sex and age) and different levels of functional independence for the elderly in their basic activities of daily living (ABVD's) such as: bathe, dress, use the bathroom for withdrawals, transfers perform, has control of the sphincters and the food itself. Subject themselves, if capable of responding to the issues of consistency index, did. The answers were given to the auxiliary nurse responsible for care to residents.
  Other Names: Elderly

SUMMARY:
Getting old is a process of transformation of the body that occurs along the vital cycle in a universal and progressive way causing functional restrictions in the human being. The aim of this work was to identify, analyze and quantify the limitations of the functional capacity of the institutionalized elderly who are not provided with physiotherapic assistance.

DETAILED DESCRIPTION:
A descriptive, qualitative, quantitative and transverse field research was made, based on an evaluation of the activities of daily living (ADL) using the Katz Index, with 62 institutionalized elderly people from Casa do Pobre de Maceió, Alagoas, both genders, average age of 77.03 years old and different levels of functions. Activities related to the self care were emphasized. At first, people were classified as independent, partially dependent and totally dependent. According to the Katz Index score, they were classified regarding their functional dependency, which varies from level 0 (a totally independent person) to level 6 (a totally dependent person in the six evaluated functions).

ELIGIBILITY:
Inclusion Criteria:

* To be elderly and a resident of Casa do Pobre de Maceió

Exclusion Criteria:

* Individuals under the age of 60 years and over 90, or received private care or physical therapy who refused to participate in the evaluation

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample, eder people.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juliana F Pontes, Principal Investigator — Centro de Estudos Superiores de Maceio
Locations (1):
- CESMAC - Centro de Estudos Superiores de Maceió, Maceió, Alagoas, Brazil